CLINICAL TRIAL: NCT07127965
Title: Exercise Adherence and Cognitive Decline: A Goal-setting and Exercise Intensity Intervention Collaboratively Developed With the Black Community
Brief Title: Exercise Adherence and Cognitive Decline: Phase 2
Acronym: MOVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Angela Bryan, Principal Investigator, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 25-0479
Record Dates: First submitted 2025-08-07; First posted 2025-08-17 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Cognitive Decline
Keywords: Goals; Goal Difficulty; Exercise Intensity; Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Moderate Intensity Exercise, Basic Goal Difficulty (Experimental): Participants are assigned to exercise at a moderate intensity and create basic goals
  Interventions: Behavioral: Goal Setting and Exercise Intensity Intervention
- Moderate Intensity Exercise, Challenging Goal Difficulty (Experimental): Participants are assigned to exercise at a moderate intensity and create challenging goals
  Interventions: Behavioral: Goal Setting and Exercise Intensity Intervention
- Vigorous Intensity Exercise, Basic Goal Difficulty (Experimental): Participants are assigned to exercise at a vigorous intensity and create basic goals
  Interventions: Behavioral: Goal Setting and Exercise Intensity Intervention
- Vigorous Intensity Exercise, Challenging Goal Difficulty (Experimental): Participants are assigned to exercise at a vigorous intensity and create challenging goals.
  Interventions: Behavioral: Goal Setting and Exercise Intensity Intervention

INTERVENTIONS:
Behavioral: Goal Setting and Exercise Intensity Intervention — Participants' goal-setting and exercise intensity are manipulated based on group assignment.

SUMMARY:
The purpose of this study is to conduct a test of a goals-based program to help people exercise more. This program was designed for individuals aged 45-65 from the Black community. Low levels of physical activity are related to health problems such as heart disease, diabetes, and cognitive decline. People of color are more negatively impacted by these conditions and have also historically been underrepresented by research seeking to increase physical activity. The investigators have developed this goals-based exercise promotion program with the help of a Black-led community-based organization (The Gyedi Project) and a Community Advisory Board made up of stakeholders in the Black community.

ELIGIBILITY:
Inclusion Criteria:

* <3 incorrect responses on the Pfeiffer Mental Status Questionnaire
* Ages 45 to 65
* Consent to be randomized to conditions
* Planning to remain in the Denver metro area for the next 14 months
* Identify as Black or African American

Exclusion Criteria:

* Currently physically active (i.e., >90 min/week of moderate PA or >40 min/week of vigorous PA consistently for the past 6 months)
* On antipsychotic medications or currently under treatment for any serious psychiatric disorder including Alzheimer's or dementia
* Inability to walk 3 blocks without chest pain, shortness of breath, or lightheadedness
* Inability to climb 2 flights of stairs without chest pain, shortness of breath, or lightheadedness

PCP Exclusion Criteria:

* Answers "yes" to 1 or more of the 7 general questions of the PAR-Q+ and answers yes to any of the follow up questions.
* Blood pressure at baseline is greater than 160/100
* Blood pressure at baseline is between 140/90 - 160/100 and the participant is currently taking blood pressure medication
* Blood pressure > 210/90 mmHg (for men) or > 190/90 mmHg (for women) immediately after exercise

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | Baseline, Visit 15 (6 Months after baseline), Visit 17 (12 months after baseline)
  Blood pressure (systolic and diastolic) of all participants is collected before the intervention
Activity Levels | Baseline, Visit 15 (6 months after baseline), Visit 17 (12 months after baseline)
  Exercise Intensity (PAR). Answers are direct (ex. how many hours active) and not scaled. Information is requested for the week and the past 3 months.
Sleep Levels | Baseline, Visit 15 (6 months after baseline), Visit 17 (12 months after followup)
  Exercise Intensity (PAR). Answers are direct (ex. how many hours did you sleep) and are not scaled. Information is requested for the past 7 days.
Exercise Intensity | Baseline, Visit 15 (6 months after baseline), Visit 17 (12 months after baseline)
  Exercise Intensity (PAR). Answers are direct (ex. how many hours did you sleep) and are not scaled. Information is requested for the past 7 days.
Exercise Behavior | Baseline, Visit 17 (12 months after Baseline)
  L-Cat. Single question that asks about frequency/rigor of physical activity, with six potential answers ranging from no physical activity to daily physical activity.
Exercise Behavior | All study timepoints (Visits 1-17; approximately 14 months)
  modified Godin Shepard Leisure Time Physical Activity Questionnaire. Measures physical and leisure activity over a typical one week period
Theoretical Mediators of Exercise Behavior | Baseline, Visit 12 (supervised exercise visit), Visits 14-17 (3, 6, 9, and 12 months after baseline)
  Intrinsic Motivation Inventory. Questions relate to how participants think or feel about physical activity, with answers ranging from 1 (strongly disagree) to 7 (strongly agree). Broader scores are broken up into subscales; final subscale scores are summed and averaged. Higher scores indicate higher agreement with that subscale.
Theoretical Mediators of Exercise Behavior | Baseline, Visit 12 (supervised exercise visit), Visits 14-17 (3, 6, 9, and 12 months after baseline)
  Self-Efficacy. 9 questions about confidence in exercise on scale of 1 (disagree strongly) to 7 (agree strongly). Higher scores indicate higher perceived confidence in doing that activity. Total scores are summed.
Theoretical Mediators of Exercise Behavior | Baseline, Visit 12 (supervised exercise visit), Visits 14-17 (3, 6, 9, and 12 months after baseline)
  Exercise Intention Survey. Scored on a Likert scale from 1 (strongly disagree) to 7 (strongly agree) to indicate level of agreement to statements related to intention to exercise. Scores are summed to produce a total score. Higher scores indicate stronger intention to exercise, lower scores indicate weaker intention.
Theoretical Mediators of Exercise Behavior | Baseline, Visit 12 (supervised exercise visit), Visits 14-17 (3, 6, 9, and 12 months after baseline)
  Exercise Identity Score. Scored on a Likert scale from 1 (strongly disagree) to 7 (strongly agree) to indicate level of agreement to statements related to attitudes towards exercise. Scores are summed and averaged to provide an overall score. Higher scores indicate a positive attitude towards exercise, lower scores less favorable attitude.
Theoretical Mediators of Exercise Behavior | Baseline, Visit 12 (supervised exercise visit), Visits 14-17 (3, 6, 9, and 12 months after baseline)
  Exercise alignment with Black identity. Assessment of the extent to which 7 common exercises are aligned with Black identity
Heart Rate Variability | Baseline, Visit 17 (12 months after Baseline)
  Heart Rate Variability is measured using chest strap monitor.
Heart Rate | Baseline, Visits 2-13 (Supervised Exercise Training, 1 hour 3x/week for 4 weeks), Visit 15 (6-month follow-up), Visit 17 (12-month follow-up)
  Heart Rate is measured using chest strap monitor.
Ventilatory Threshold | Baseline
  Talk Test. Graded treadmill test where intensity is increased at intervals to determine participant's ventilatory threshold.
Perceived Exertion | Baseline, Visits 2-13 (Supervised Exercise Training, 1 hour 3x/week for 4 weeks)
  A single-item measure from Borg (1973) was used to assess participants' rate of perceived exertion (RPE) during the exercise bout. Participants were asked to rate the average intensity of exercise [at that moment/during the past ten minutes] on a 25-point scale ranging from 6 (no exertion at all) to 20 (maximal exertion).
Pain Levels | Visits 2, 6, 12 (Supervised Exercise Training)
  A single item measure from Borg (1998) was used to assess participants' pain levels during the exercise bout. Participants were asked to indicate how much pain they felt [at that moment/during the past ten minutes] on an 11-point scale ranging from 0 (nothing at all) to 10 (excruciating).
Affective Valence | Visit 12, Visits 14-16 (3, 6, and 9 months after baseline)
  The Feeling Scale, a single-item measure from Hardy and Rejeski (1989), was used to assess participants' affective valence during the exercise bout. Participants were asked to indicate how they felt [at that moment/during the past ten minutes] on an 11-point scale ranging from -5 (very bad) to +5 (very good).
Affective Arousal | Visits 2, 6, 12 (Supervised Exercise Training)
  The Felt Arousal Scale, a single-item measure from Svebak and Murgatroyd (1985), was used to assess participants' affective arousal during the exercise bout. Participants were asked to indicate how "worked-up" they felt [at that moment/during the past ten minutes] on a 6-point scale ranging from 1 (low arousal) to 6 (high arousal).
Enjoyment | Visits 2, 6, 12 (Supervised Exercise Training)
  A single item measure from Gillman and Bryan (2015) was used to assess participants' enjoyment levels during the exercise bout. Participants were asked to indicate how enjoyable exercise was [at that moment/during the past ten minutes] on a 5-point scale ranging from 1 (no enjoyment at all) to 5 (a great deal of enjoyment).
Exercise Check-In | Visits 14-17 (3, 6, 9, and 12 months after baseline)
  Three short questions assessing if the participant planned to engage in exercise and how many minutes of moderate (0-120) and vigorous (0-60) exercise they engaged in
Exercise Benefits and Barriers | Baseline, Visit 12 (supervised exercise visit), Visits 14-17 (3, 6, 9, and 12 months after baseline)
  A 10 item scale assessing perceived benefits of and barriers to exercise
Anthropometrics | Baseline, Visit 17 (12-month follow-up)
  Height will be measured in centimeters
Diet | Baseline, Visit 17 (12-month follow-up)
  NCI's Eating at America's Table Study (EATS) Fruit & Vegetable All-Day Screener. A short dietary assessment instrument for measuring fruit and vegetable intake over the past month.
Demographics | Baseline
  Survey includes gender, sexual orientation, age, detailed race/ethnicity, and SES
Objective Physical Activity | Baseline, Visit 15 (6 months after baseline), Visit 17 (12 months after baseline)
  Objective physical activity will be measured through ActiGraph. Participants will be given the ActiGraph at baseline and will be asked to wear the device for one week. Participants will then be asked to wear the watch continuously for the week before visit 15 (6-month follow-up) and visit 17 (12-month follow-up).
Biomarkers of Cognitive Aging | Baseline and Visit 17 (12 months after baseline)
  Biomarkers of cognitive again will be analyzed by blood samples. Blood samples will be collected at baseline and Visit 17 (12-month follow-up) and stored. At the end of the study, samples will be sent for analysis of biomarkers involved in cognitive aging, including p-tau181, NfL, Ab40, Ab42, GFAP, and IGF-1.
Anthropometrics | Baseline, Visit 17 (12-month follow-up)
  Weight will be measured in pounds

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Recreation Centers in the Denver Metro Area, Aurora, Colorado
  - University of Colorado at Boulder, Boulder, Colorado